CLINICAL TRIAL: NCT06005636
Title: Risk Factors and Risk Prediction Model for Post-stroke Delirium in Ischemic Stroke Patients
Brief Title: Post-stroke Delirium in Ischemic Stroke Patients
Status: Completed | Type: Observational
Sponsor: Jinan University Guangzhou (Other)
Collaborators: First Affiliated Hospital of Jinan University (Other)
Responsible Party: Principal Investigator, Xiaoyan Cai, Ms, Jinan University Guangzhou
Other Study IDs: KY-2021-106
Record Dates: First submitted 2023-08-17; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- with post-stroke delirium: ischemic stroke patients with post-stroke delirium
  Interventions: Diagnostic Test: Test delirium state
- without post-stroke delirium: ischemic stroke patients without post-stroke delirium
  Interventions: Diagnostic Test: Test delirium state

INTERVENTIONS:
Diagnostic Test: Test delirium state — use scale to test whether ischemic stroke patients have post-stroke delirium

SUMMARY:
This study is to investigate the predictors of post-stroke delirium, develop and validate a nomogram of post-stroke delirium in the ischemic stroke patients.

DETAILED DESCRIPTION:
Introduction: Post-stroke delirium (PSD) is associated with unfavorable prognosis. Effectively identifying risk factors of PSD and predicting PSD is of essential.

Methods: This is a prospective, single-centered, cohort study.

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥18 years old;(2) ischemic stroke, confirmed by computed tomography (CT) or magnetic resonance imaging (MRI) scans;(3) patients or their agencies agree to participate in this study.

Exclusion Criteria:

1. brain dysfunction caused by non-vascular causes such as traumatic brain injury, brain tumor or metastatic brain tumor;(2) history of serious mental illness such as schizophrenia;(3) unable to cooperate to the assessment as deafness, blindness, aphasia, dysarthria;(4) be in coma [Glasgow Coma Scale (GCS)≤8 points] or sedation [Richmond Agitation Sedation Scale (RASS)<-3 points], and do not ameliorate during study;(5) with incomplete data.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ischemic stroke patients were recruited from a Grade 3A hospital in Southern China.
Sampling Method: Non-Probability Sample
Enrollment: 985 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-10 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
post-stroke delirium | The first week of admission

CONTACTS AND LOCATIONS:
Overall Officials: Fengxia Yan, Principal Investigator — Jinan University
Locations (1):
- the First Affiliated Hospital of Jinan University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No